CLINICAL TRIAL: NCT03052894
Title: Validation of a Device to Monitor Muscle Relaxation During Surgery
Brief Title: Validation of a Muscle Relaxation Monitor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection issues from the electronic health record.
Sponsor: Richard H Epstein (Other)
Collaborators: Society for Technology in Anesthesia (Unknown); University of Miami (Other)
Responsible Party: Sponsor-Investigator, Richard H Epstein, Professor of Clinical Anesthesiology, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20161018
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Neuromuscular Blockade
Keywords: anesthesiology; neuromuscular blockade; monitoring device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hydraulic Monitoring Device (Experimental): Monitoring device to be compared to electromyographic (EMG) device in the same patient; measures depth of neuromuscular blockade during general anesthesia based on the pressure exerted by the muscles of the thumb.
  Interventions: Device: Hydraulic Monitoring Device
- Standard EMG Monitoring Device (Active Comparator): Currently used standard monitoring device; measures depth of neuromuscular blockade during general anesthesia based on the action potential of the muscles of the thumb.
  Interventions: Device: Standard EMG Monitoring Device

INTERVENTIONS:
Device: Hydraulic Monitoring Device — The hydraulic monitoring device externally measures the pressure associated with thumb strength applied to the device to determine the depth of neuromuscular blockade during general anesthesia.
  This will be compared to measurements using a current monitoring device in the same patient.
  Arms: Hydraulic Monitoring Device
Device: Standard EMG Monitoring Device — Standard and in current usage, the electromyographic monitoring (EMG) device externally measures the action potential of the muscles of the thumb to determine the depth of neuromuscular blockade during general anesthesia.
  This will be used as the clinical monitoring device and as a comparator.
  Arms: Standard EMG Monitoring Device

SUMMARY:
The objective of this study is to determine the accuracy of a hydraulically coupled twitch monitor compared to the EMG twitch monitor in current use to measure the extent of neuromuscular blockade in patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Neuromuscular blockade (paralysis) is necessary for many surgical procedures to provide optimal surgical conditions. The extent of paralysis typically assessed during routine clinical care by examining the muscle response of the thumb ("twitch") following delivery of a series of the "train-of-four".

Quantitative assessment of neuromuscular block can be assessed using electromyography (EMG) This technique measures action potential in the muscles of the thumb.

The proposed method is a simple technique that can constructed with equipment that is readily available in most operating rooms. If validated, it would provide a simple method to assess quantitatively the extent of neuromuscular blockade and recovery of muscle strength.

ELIGIBILITY:
1. Age >18
2. Surgery is elective
3. Subject has been NPO for fluids for >2 hours and for solids >8 hours
4. General anesthesia with tracheal intubation is required
5. Mask ventilation is expected to be without difficulty
6. Subject voluntarily consents in writing to the protocol
7. ASA Physical Status 1-III (healthy individuals, those with mild comorbid conditions, or those with more serious co-morbid conditions that are well controlled)

Exclusion Criteria:

1. Lack of ability to provide written, informed consent
2. Airway examination indicates a likelihood of difficult mask ventilation
3. Symptoms of active reflux at the time of induction, at risk of having food in their stomach at the time of induction, expected abnormal response to non-depolarizing neuromuscular blockers
4. Age ≤18 years
5. Pregnant women
6. Presence of carpal tunnel syndrome
7. Prisoners
8. General anesthesia not being provided
9. Tracheal intubation will not be performed
10. Anticipated length of surgery <60 minutes
11. Emergent or urgent surgery
12. Disease that might alter the normal neuromuscular response to electrical stimulation (e.g., muscular dystrophies, myasthenia gravis, quadriplegia).
13. ASA Physical Status IV or V (individuals with major comorbid conditions that are a constant source of risk to health)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Hydraulic Twitch Monitoring Device in Measuring Neuromuscular Blockade as Compared to EMG Monitoring Device, Assessed using Repeated Measures Bland-Altman Analysis | 12 months
  To determine the accuracy (bias and precision) of a the monitoring device as compared to the electromyographic (EMG) monitor in measuring the extent of neuromuscular blockade in subjects undergoing general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Epstein, MD, Principal Investigator — University of Miami
Locations (1):
- Department of Anesthesiology at University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brull SJ, Silverman DG. Visual assessment of train-of-four and double burst-induced fade at submaximal stimulating currents. Anesth Analg. 1991 Nov;73(5):627-32. doi: 10.1213/00000539-199111000-00020. PMID 1952146
- [Result] Viby-Mogensen J, Jensen NH, Engbaek J, Ording H, Skovgaard LT, Chraemmer-Jorgensen B. Tactile and visual evaluation of the response to train-of-four nerve stimulation. Anesthesiology. 1985 Oct;63(4):440-3. doi: 10.1097/00000542-198510000-00015. No abstract available. PMID 4037404
- [Result] Brull SJ, Murphy GS. Residual neuromuscular block: lessons unlearned. Part II: methods to reduce the risk of residual weakness. Anesth Analg. 2010 Jul;111(1):129-40. doi: 10.1213/ANE.0b013e3181da8312. Epub 2010 May 4. PMID 20442261
- [Result] Ali HH, Utting JE, Gray TC. Quantitative assessment of residual antidepolarizing block. II. Br J Anaesth. 1971 May;43(5):478-85. doi: 10.1093/bja/43.5.478. No abstract available. PMID 4254032
- [Result] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Result] Kopman AF, Yee PS, Neuman GG. Relationship of the train-of-four fade ratio to clinical signs and symptoms of residual paralysis in awake volunteers. Anesthesiology. 1997 Apr;86(4):765-71. doi: 10.1097/00000542-199704000-00005. PMID 9105219
- [Result] Eriksson LI, Sundman E, Olsson R, Nilsson L, Witt H, Ekberg O, Kuylenstierna R. Functional assessment of the pharynx at rest and during swallowing in partially paralyzed humans: simultaneous videomanometry and mechanomyography of awake human volunteers. Anesthesiology. 1997 Nov;87(5):1035-43. doi: 10.1097/00000542-199711000-00005. PMID 9366453
- [Result] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929